CLINICAL TRIAL: NCT02002286
Title: Pilot Study: Safety and Efficacy Study of Tripterygium Wilfordii Hook F Extract in cART-Treated HIV Patients With Poor Immune Responses
Brief Title: Safety and Efficacy Study of TwHF in HIV Patients With Poor Immune Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LI Taisheng (Other)
Responsible Party: Sponsor-Investigator, LI Taisheng, Professor, Peking Union Medical College
Organization: Peking Union Medical College (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TwHF Pilot
Record Dates: First submitted 2013-11-18; First posted 2013-12-05 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-11

CONDITIONS: HIV
Keywords: HIV-infected immunological non-responders; Tripterygium Wilfordii Hook F; Immune activation
MeSH Terms: interventions — Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TwHF extract + cART (Experimental): Use Tripterygium Wilfordii Hook F extract (TwHF extract) and continue current cART regimen
  Interventions: Drug: Tripterygium Wilfordii Hook F extract (TwHF extract); Drug: cART
- cART control (Other): Continue current cART regimen
  Interventions: Drug: cART

INTERVENTIONS:
Drug: Tripterygium Wilfordii Hook F extract (TwHF extract) — The extract Tripterygium wilfordii Hook F (TwHF), a traditional Chinese medication, has been used as anti-inflammatory therapy to treat autoimmune diseases including rheumatoid arthritis and Crohn's disease.
  Other Names: Triptolide Wilfordii
  Arms: TwHF extract + cART
Drug: cART — Participants who will be enrolled in this trial would keep their previous combined antiretroviral therapy, such as zidovudine or stavudine plus lamivudine plus nevirapine or efavirenz.
  Other Names: Combination antiretroviral therapy

SUMMARY:
This study is a pilot study to evaluate impact of Tripterygium Wilfordii Hook F (TwHF) on T cell immune activation and immune activation in HIV-infected immunological non-responders. The investigators aim to evaluate the safety and efficacy profiles of TwHF in HIV immunological non-responders.

DETAILED DESCRIPTION:
The investigators recruited 23 patients from Peking Union Medical College Hospital Outpatient clinic. They were all immunological non-responders. Nineteen patients will receive Triptolide wilfordii Hook F extract (10mg tid po) plus current cART, while 4 patients will continue their current cART. This study will last for 12 months. Patients will be followed up at month 0, 3, 6, 9, and 12. During each follow-up time point, adverse effects, T cell subsets, T cell activation markers and other routine tests will be ordered. The investigators hypothesis that TwHF might boost CD4 cell recovery by reducing immune activation.

ELIGIBILITY:
Inclusion Criteria:

* Continuous antiretroviral therapy > 18 months, and consistent HIV-RNA< 40 copies/mL more than 12 months;
* 18-65 years old;
* Male or female;
* Good adherence and promise to follow-up;
* Inform Consent signed;
* CD4 T cells less than 300/ul .

Exclusion Criteria:

* Active opportunistic infection (not stable within 4 weeks 2 weeks ) or AIDS-related carcinoma;
* Hemoglobin (HGB) < 9 g/dl, white blood cell (WBC) < 2000/ul, granulin (GRN) < 1000 /ul, platelet (PLT) < 75000 /ul, Cr >1.5x ULN, ALT or AST or alkaline phosphatase (ALP) >3x upper limit of normal (ULN), total bilirubin (TBIL) >2x ULN, creatine kinase (CK) > 2x ULN;
* Pregnant or breastfeeding woman or woman with pregnancy plan;
* Active drug-user;
* Severe neurological defects;
* Active alcohol abuse;
* Severe gastrointestinal ulcer .
* End-stage disease such as cirrhosis, chronic obstructive pulmonary disease, congestive heart failure, recent myocardial ischemia,tumor, etc Those who are undertaking steroids, immunomodulator, anti-inflammatory agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Changes of T cell subsets and immune activation markers | 12 months
  T cell subsets and activation biomarkers including CD4 count, memory and naive CD4 cell count, and CD38/HLA-DR expression will be monitored.

SECONDARY OUTCOMES:
Viral load | 12 months
  During follow-up, viral load will also be monitored.
Number of participants with adverse events as a measure of safety and tolerability | 12 months
  During each follow-up time point, clinical status and adverse effects will also be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Taisheng Li, MD, PhD, Principal Investigator — Department of Infectious Diseases, Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- [Background] Piconi S, Parisotto S, Rizzardini G, Passerini S, Terzi R, Argenteri B, Meraviglia P, Capetti A, Biasin M, Trabattoni D, Clerici M. Hydroxychloroquine drastically reduces immune activation in HIV-infected, antiretroviral therapy-treated immunologic nonresponders. Blood. 2011 Sep 22;118(12):3263-72. doi: 10.1182/blood-2011-01-329060. Epub 2011 May 16. PMID 21576701
- [Background] Murray SM, Down CM, Boulware DR, Stauffer WM, Cavert WP, Schacker TW, Brenchley JM, Douek DC. Reduction of immune activation with chloroquine therapy during chronic HIV infection. J Virol. 2010 Nov;84(22):12082-6. doi: 10.1128/JVI.01466-10. Epub 2010 Sep 15. PMID 20844049
- [Derived] Li T, Xie J, Li Y, Routy JP, Li Y, Han Y, Qiu Z, Lv W, Song X, Sun M, Zhang X, Wang F, Jiang H. Tripterygium wilfordii Hook F extract in cART-treated HIV patients with poor immune response: a pilot study to assess its immunomodulatory effects and safety. HIV Clin Trials. 2015 Mar-Apr;16(2):49-56. doi: 10.1179/1528433614Z.0000000005. Epub 2015 Jan 26. PMID 25874991